CLINICAL TRIAL: NCT05209373
Title: Compassionate And Loving Mindset Towards HEART Health riSk (CALM HEARTS 2): A Randomized Optimization Trial
Brief Title: Optimizing a Self-compassion Intervention Designed to Improve Physical Activity Among Women at Risk for Heart Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HE2021-0175
Record Dates: First submitted 2022-01-10; First posted 2022-01-26 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Cardiovascular Diseases
Keywords: self-compassion; physical activity; self-regulation; randomized optimization trial; emotions
MeSH Terms: conditions — Cardiovascular Diseases; Motor Activity; Self-Control

STUDY DESIGN:
Masking Description: A third-party with no involvement in intervention delivery or data analysis will use a random numbers list generated by the IBM Statistical Package for the Social Sciences (SPSS) 28© (statistical software) to allocate participants to the two intervention conditions. The random number list will not be accessible to research staff involved in recruitment and intervention delivery. The results of allocation will not be revealed until participants begin the intervention sessions in their respective conditions.
  Complete blinding of facilitators and participants is not possible; facilitators and participants will know if they are in the individual or group condition but will be blind to participants' pre-intervention self-compassion score.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group-Delivered Self-Compassion Intervention (Experimental): A 4-week intervention pairing behaviour change and self-compassion education, aimed to increase physical activity and help women cope with their risk of cardiovascular disease. Participants in the group condition will complete Sessions 2-4 with 6-9 other participants plus a facilitator. Both conditions will be exposed to identical intervention content. All intervention sessions will be hosted on an institution-sponsored Zoom videoconferencing account.
  Week 1, Session 1 (60 minutes): Participants will meet in their group to discuss CVD risk factors and set physical activity goals.
  Weeks 2-4, Sessions 2-4 (60 minutes each): Participants will meet in their group to receive self-compassion education to aimed at encouraging adaptive coping with cardiovascular risk and physical activity behaviour change. Brief self-compassionate writing exercises will be assigned as home practice after Sessions 2-4.
  Interventions: Behavioral: Intervention Condition
- Positive control condition: Individually-Delivered Self-Compassion Intervention (Other): A 4-week intervention pairing behaviour change and self-compassion education, aimed to increase physical activity and help women cope with their risk of cardiovascular disease. Participants in the individual condition will complete Sessions 2-4 individually with a facilitator. Both conditions will be exposed to identical intervention content. All intervention sessions will be hosted on an institution-sponsored Zoom videoconferencing account.
  Week 1, Session 1 (60 minutes): Participants will meet individually with a facilitator to discuss CVD risk factors and set physical activity goals.
  Weeks 2-4, Sessions 2-4 (60 minutes each): Participants will meet individually with a facilitator to receive self-compassion education to aimed at encouraging adaptive coping with cardiovascular risk and physical activity behaviour change. Brief self-compassionate writing exercises will be assigned as home practice after Sessions 2-4.
  Interventions: Behavioral: Positive Control Condition

INTERVENTIONS:
Behavioral: Intervention Condition — 4-week intervention combining behaviour change and self-compassion education to promote coping with CVD risk and increased engagement in physical activity.
  Arms: Group-Delivered Self-Compassion Intervention
Behavioral: Positive Control Condition — 4-week intervention combining behaviour change and self-compassion education to promote coping with CVD risk and increased engagement in physical activity.
  Arms: Positive control condition: Individually-Delivered Self-Compassion Intervention

SUMMARY:
The investigators aim to optimize an intervention which teaches women at risk for cardiovascular disease (CVD) to cope with this risk using self-compassion (an attitude of kindness towards oneself) in order to adopt a physically active lifestyle.

The investigators previously conducted a one-on-one self-compassion intervention for 11 women with CVD risk that successfully increased physical activity. However, meeting one-on-one with each participant was time and resource intensive.

The primary purpose of the present study is to determine if group self-compassion intervention delivery is comparably effective to one-on-one delivery for increasing physical activity among women at risk for CVD. The investigators hypothesize that group delivery should be at least as effective as individual delivery at increasing physical activity.

Furthermore, only women low in self-compassion were included in the previous study. The secondary purpose of the present study is to determine if women higher in self-compassion can also benefit from the intervention. The investigators hypothesize that participants at all levels of self-compassion should benefit similarly from the intervention.

Finally, the tertiary purpose is to determine if delivery mode and self-compassion interact such that one method of delivery (group or one-on-one) is better suited to women at low, moderate, or high self-compassion. This outcome is exploratory only and the researchers present no hypothesis.

The present study follows the methods of a randomized optimization trial. Women at risk for CVD will be randomly assigned to receive four sessions of combined physical activity behaviour change and self-compassion training in groups of six to nine or through one-on-one delivery. The intervention will provide one session to discuss participants' CVD risk and physical activity goals, and then three sessions of self-compassion training.

Outcome measures will be assessed pre- and post-intervention. The effectiveness of the one-on-one and group conditions for improving the study outcomes will be examined. The present research will determine how best to deliver an intervention which teaches women to cope with their CVD risk using self-compassion in order to become more physically active. The results of the present study will inform an eventual efficacy trial.

DETAILED DESCRIPTION:
In preparation for the proposed research, the investigators conducted a one-arm pilot intervention (N=11) to examine the feasibility and acceptability of a self-compassion intervention for women at risk for cardiovascular disease (CVD). This pilot study established proof-of-concept (Czajkowski et al., 2015) for this intervention by producing a clinically significant increase in physical activity (M=837.5 Metabolic Equivalent (MET)*minutes per week; Florido et al., 2018). Further, feasibility criteria for recruitment time (1 week), retention rate (100%), and completion of study measures (97%) successfully exceeded the pre-established standards. Exit surveys found the intervention was 100% acceptable to participants. These results are encouraging yet questions remain about how best to deliver the intervention and with whom.

An optimization trial is the appropriate iterative step that will refine the present feasible and acceptable intervention with established proof of concept prior to conducting an efficacy trial. The present optimization trial will advance a research program informed by The ORBIT Model for Behavioural Treatment Development (Czajkowski et al., 2015). Two identified shortcomings of the pilot intervention will be targeted for optimization.

Primary Optimization Target: The pilot intervention was delivered individually to each participant. For 11 participants to complete the study, 33 individual meetings totalling over 40 hours were required over three weeks. This resource intensive delivery method may not be practical. Delivering the intervention to small groups would be more practical. Therefore, the primary objective of this optimization trial is to determine if a self-compassion intervention delivered in small groups is at least as effective at increasing physical activity among women at risk for CVD compared to a self-compassion intervention delivered individually. The investigators hypothesize that group delivery should be at least as effective as individual delivery at increasing physical activity.

Secondary Optimization Target: The previous pilot intervention only included women with CVD risk who were low on self-compassion. While women low on self-compassion are an obvious intervention target, women with moderate or high self-compassion may also benefit from learning to apply their self-compassion to their CVD risk and physical activity efforts. No research exists to inform the effectiveness of self-compassion interventions when delivered to participants low, moderate, and high on self-compassion. Therefore, the secondary objective of this optimization trial is to determine if baseline self-compassion influences physical activity, behavioural outcomes, or psychological outcomes of the intervention. The investigators hypothesize that participants at all levels of self-compassion should benefit similarly from the intervention. Finally, the tertiary objective is to determine if delivery mode and self-compassion interact such that one method of delivery (group or individual) is better suited to women at low, moderate, or high self-compassion. This outcome is exploratory only and the researchers put forth no hypothesis.

Trial Design: This intervention was developed with the Consolidated Standards of Reporting Trials (CONSORT) guidelines (Schulz et al., 2010). This is a two-armed optimization trial with 1:1 randomization to be conducted in a single centre in Manitoba, Canada. Women at risk for CVD will be randomized to receive a combined physical activity behaviour change plus self-compassion intervention in small groups (intervention condition) or individually with a facilitator (control condition). The individual condition serves as a positive control against which the effectiveness of the group condition at increasing physical activity will be judged. The intervention will be delivered to both conditions via an institution-sponsored videoconferencing platform. Data will be collected at pre- and post-intervention using validated surveys completed online. The investigators often use this data collection approach.

Participants: Participants will be women at risk for CVD identified through the Women's Advanced Risk-assessment in Manitoba (WARM) Hearts Cohort (NCT03938155), a large, ongoing prospective study to improve CVD risk detection in Manitoban women. Participants identified through pre-screening will be contacted by telephone and invited to participate in the study. Interested individuals will be sent an online questionnaire by email to assess the study eligibility criteria. Eligible individuals will be stratified by self-compassion score and sampled to equally enroll participants scoring low, moderate, and high on self-compassion. This recruitment strategy is required for the planned method of statistical analysis.

Randomization: Participants will be randomly allocated to the two intervention conditions with a 1:1 ratio. The random number list will not be accessible to research staff involved in recruitment and intervention delivery. The results of allocation will not be revealed until participants begin the intervention sessions in their respective conditions.

Intervention: Participants will engage in four, weekly one-hour sessions delivered by research assistants trained in self-compassion (six-week course). Both facilitators will deliver interventions to a similar number of participants in both conditions by alternating between conditions every four weeks. Intervention delivery will be guided by a script to prevent drift. To ensure facilitator fidelity, 20% of all intervention sessions will be recorded and shared with a self-compassion expert for feedback. This intervention draws from the Mindful Self-Compassion Program (Neff & Germer, 2013) and was developed by self-compassion experts.

Participants in the group condition will complete the four weekly sessions with six to nine other participants plus a facilitator; those in the individual condition will meet individually with a facilitator. Both conditions will be exposed to identical intervention content.

In Session One participants will discuss risk factors for CVD, be advised of the Canadian 24-Hour Movement Guidelines (Ross et al., 2020) and guided to set a physical activity goal using the SMART goals framework (American College of Sports Medicine, 2017).

In Session Two, participants will apply the three components of self-compassion (self-kindness, mindfulness, and common humanity) (Neff, 2003) to their CVD risk and physical activity efforts.

In Session Three, participants will learn to use the Yin (gentle; Neff, 2003) side of self-compassion to cope with difficult emotions, and the Yang (fierce, Neff, 2003) side of self-compassion to improve their health through physical activity.

In Session Four, participants will use the mindful practices of savouring and gratitude (Neff, 2003) to find enjoyment in physical activity.

Identical self-compassion writing exercises will be assigned to both conditions as home practice after Sessions 2-4.

Outcomes: Reliable and valid measures will be distributed using SurveyMonkey (www.momentive.ai) at pre-intervention and post-intervention.

Statistics: The sample required to achieve statistical power is 82 participants. The power analysis was conducted based on data showing that 10-minute increases in daily moderate to vigorous physical activity significantly lower CVD risk (Glazer et al., 2013). To protect against approximately 15% attrition (Ferrari et al., 2019) 96 participants will be enrolled in the trial.

Analyses will employ a 2 by 3 factorial ANOVA to address the three study objectives. Each factor in a factorial ANOVA is controlled for within the combinations of factors tested. The primary objective of the study is to determine if the group condition (intervention condition) is at least as effective as the individual condition (control condition) at increasing physical activity. The factorial ANOVA will test for main effects of the group condition on post-intervention physical activity across all levels of self-compassion, controlling for effects of the individual condition. The secondary and tertiary objectives of this study are to determine if baseline self-compassion influences how women respond to the intervention, and if delivery method and self-compassion interact such that one method of delivery is better suited to women higher or lower in self-compassion. The factorial ANOVA will explore main and interaction effects between baseline self-compassion (low, moderate, high) and intervention condition (group or individual) on physical activity, behavioural outcomes, and psychological outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age 55 years or older
* Flagged response on CANHEART Index (Maclagan et al., 2014) (response of "yes" to having high blood pressure)
* Insufficient self-reported physical activity relative to guidelines of 150 minutes of moderate to vigorous physical activity per week.
* No current or planned enrolment in programming similar to the intervention
* No current diagnosis of cardiovascular disease
* No medical conditions that make it unsafe to engage in physical activity
* Available for all intervention sessions
* Comfortable using videoconferencing
* Comfortable reading and communicating in English

Score on the self-compassion scale will be monitored in order to ensure equal enrolment of participants scoring low, moderate, and high on the self-compassion scale (Neff, 2021). Eligibility criteria may be adjusted according to self-compassion score in order to represent the full range of possible self-compassion scores.

Exclusion Criteria:

* Being under 50 years old
* No flagged response on CANHEART Index (Maclagan et al., 2014) (response of "no" to having high blood pressure)
* Self-report meeting or exceeding guidelines of 150 minutes of moderate to vigorous physical activity per week.
* Current or planned enrolment in programming similar to the intervention
* Current diagnosis of cardiovascular disease
* Medical conditions that make it unsafe to engage in physical activity
* Not available for all intervention sessions
* Not comfortable using videoconferencing
* No comfortable reading and communicating in English

Min Age: 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2022-01-09 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Differences between groups in moderate to vigorous physical activity from pre-intervention to post-intervention | Post-intervention (4 week time point)
  International Physical Activity Questionnaire (Craig et al., 2003). Seven items to measure frequency and duration of weekly walking, moderate physical activity, and vigorous physical activity, and sitting.

SECONDARY OUTCOMES:
Differences between groups in self-compassion from pre-intervention to post-intervention | Post-intervention (4 week time point)
  The Self-Compassion Scale (Neff, 2003a); this 26-item scale assesses current level of compassion for oneself. The scale has 6 sub-scales (self-kindness, self-judgment, mindfulness, over-identification, isolation, common humanity. Participants use a 5-point Likert scale ranging from 1 (almost never) to 5 (almost always) to provide responses. The six sub-scale means are first calculated and then a total self-compassion score is calculated using the overall mean of the sub scales.
Differences between groups in general health promoting behaviours from pre-intervention to post-intervention | Post-intervention (4 week time point)
  Health Promoting Lifestyle Profile II (Walker et al., 1995); this 52 item scale assesses current engagement in health promoting behaviours. This scale has six sub-scales (physical activity, health responsibility, nutrition, spiritual growth, interpersonal relations, stress management). Participants respond using a 4-point Likert scale ranging from 1 (never) to 4 (routinely). The six sub-scale means are first calculated and then a total health-promoting behaviour score is calculated using the overall mean of the sub scales.
Differences between groups in health anxiety and illness self-blame from pre-intervention to post-intervention | Post-intervention (4 week time point)
  Two subscales of the Multidimensional Health Questionnaire (MHQ; Snell & Johnson, 1997) will be used to assess health anxiety and illness self-blame. Each sub-scale uses five items to assess its respective outcome. Participants indicate their level of agreement with each statement using a 5-point Likert scale ranging from 1 (not at all characteristic of me) to 5 (very characteristic of me). Means are calculated from the items of each sub-scale to calculate Health Anxiety and Illness Self-Blame
Differences between groups in health behaviour intentions from pre-intervention to post-intervention | Post-intervention (4 week time point)
  Participants will respond to six items assessing their intentions to engage in health promoting behaviours over the next month. Intentions assessed include physical activity, healthy eating, seeking advice of a medical professional, smoking cessation (if applicable), weight reduction (if applicable), and inquiry about healthy living resources. Similar methods have been used by Semenchuk et al., (2020). Participants respond to each item using a 7-point Likert scale ranging from 1 (strongly disagree) to 7 (strongly agree). Descriptive statistics are then reported to examine which behaviours participants intended to change, the strength of these subjective intentions.
Personal Growth Initiative as a potential mediator | Post-intervention (4 week time point)
  Personal Growth Initiative Scale-II (Robitschek et al., 2012); This 16-item scale assesses four dimensions of personal growth initiative: Readiness for Change, Planfulness, Using Resources, and Intentional Behaviour. Participants rate their agreement with each item using a 6-point likert scale ranging from 0 (disagree strongly) to 5 (agree strongly). Mean scores are calculated for each sub-scale, then a grand mean Personal Growth Initiative score is calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Manitoba, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Collins LM, Dziak JJ, Kugler KC, Trail JB. Factorial experiments: efficient tools for evaluation of intervention components. Am J Prev Med. 2014 Oct;47(4):498-504. doi: 10.1016/j.amepre.2014.06.021. Epub 2014 Aug 1. PMID 25092122
- [Background] American College of Sports Medicine. ACSM Guidelines for Exercise Testing and Prescription. 10th ed. London: Wolters Kluwer; 2017.
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Czajkowski SM, Powell LH, Adler N, Naar-King S, Reynolds KD, Hunter CM, Laraia B, Olster DH, Perna FM, Peterson JC, Epel E, Boyington JE, Charlson ME. From ideas to efficacy: The ORBIT model for developing behavioral treatments for chronic diseases. Health Psychol. 2015 Oct;34(10):971-82. doi: 10.1037/hea0000161. Epub 2015 Feb 2. PMID 25642841
- [Background] Ferrari, M., Hunt, C., Harrysunker, A., Abbott, M. J., Beath, A. P., & Einstein, D. A. (2019). Self-Compassion Interventions and Psychosocial Outcomes: a Meta-Analysis of RCTs. Mindfulness, 10(8), 1455-1473. https://doi.org/10.1007/s12671-019-01134-6
- [Background] Florido R, Kwak L, Lazo M, Nambi V, Ahmed HM, Hegde SM, Gerstenblith G, Blumenthal RS, Ballantyne CM, Selvin E, Folsom AR, Coresh J, Ndumele CE. Six-Year Changes in Physical Activity and the Risk of Incident Heart Failure: ARIC Study. Circulation. 2018 May 15;137(20):2142-2151. doi: 10.1161/CIRCULATIONAHA.117.030226. Epub 2018 Jan 31. PMID 29386202
- [Background] Glazer NL, Lyass A, Esliger DW, Blease SJ, Freedson PS, Massaro JM, Murabito JM, Vasan RS. Sustained and shorter bouts of physical activity are related to cardiovascular health. Med Sci Sports Exerc. 2013 Jan;45(1):109-15. doi: 10.1249/MSS.0b013e31826beae5. PMID 22895372
- [Background] Maclagan LC, Park J, Sanmartin C, Mathur KR, Roth D, Manuel DG, Gershon A, Booth GL, Bhatia S, Atzema CL, Tu JV. The CANHEART health index: a tool for monitoring the cardiovascular health of the Canadian population. CMAJ. 2014 Feb 18;186(3):180-7. doi: 10.1503/cmaj.131358. Epub 2013 Dec 23. PMID 24366893
- [Background] Neff, K. D. (2003). The Development and Validation of a Scale to Measure Self-Compassion. Self and Identity, 2(3), 223-250. https://doi.org/10.1080/15298860309027
- [Background] Neff KD, Germer CK. A pilot study and randomized controlled trial of the mindful self-compassion program. J Clin Psychol. 2013 Jan;69(1):28-44. doi: 10.1002/jclp.21923. Epub 2012 Oct 15. PMID 23070875
- [Background] Neff, K. D., Tóth-Király, I., Knox, M. C., Kuchar, A., & Davidson, O. (2021). The Development and Validation of the State Self-Compassion Scale (Long- and Short Form). Mindfulness, 12(1). https://doi.org/10.1007/s12671-020-01505-4
- [Background] Robitschek C, Ashton MW, Spering CC, Geiger N, Byers D, Schotts GC, Thoen MA. Development and psychometric evaluation of the Personal Growth Initiative Scale-II. J Couns Psychol. 2012 Apr;59(2):274-87. doi: 10.1037/a0027310. Epub 2012 Feb 20. PMID 22352950
- [Background] Ross R, Chaput JP, Giangregorio LM, Janssen I, Saunders TJ, Kho ME, Poitras VJ, Tomasone JR, El-Kotob R, McLaughlin EC, Duggan M, Carrier J, Carson V, Chastin SF, Latimer-Cheung AE, Chulak-Bozzer T, Faulkner G, Flood SM, Gazendam MK, Healy GN, Katzmarzyk PT, Kennedy W, Lane KN, Lorbergs A, Maclaren K, Marr S, Powell KE, Rhodes RE, Ross-White A, Welsh F, Willumsen J, Tremblay MS. Canadian 24-Hour Movement Guidelines for Adults aged 18-64 years and Adults aged 65 years or older: an integration of physical activity, sedentary behaviour, and sleep. Appl Physiol Nutr Metab. 2020 Oct;45(10 (Suppl. 2)):S57-S102. doi: 10.1139/apnm-2020-0467. PMID 33054332
- [Background] Schulz KF, Altman DG, Moher D; CONSORT Group. CONSORT 2010 statement: updated guidelines for reporting parallel group randomised trials. BMJ. 2010 Mar 23;340:c332. doi: 10.1136/bmj.c332. PMID 20332509
- [Background] Semenchuk BN, Boreskie KF, Hay JL, Miller C, Duhamel TA, Strachan SM. Self-compassion and responses to health information in middle-aged and older women: An observational cohort study. J Health Psychol. 2021 Oct;26(12):2231-2247. doi: 10.1177/1359105320909860. Epub 2020 Mar 7. PMID 32148104
- [Background] Snell, W. E., & Johnson, G. (1997). The Multidimensional Health Questionnaire. American Journal of Health Behavior, 21(1), 33-42.
- [Background] Walker SN, Sechrist KR, Pender NJ. The Health-Promoting Lifestyle Profile: development and psychometric characteristics. Nurs Res. 1987 Mar-Apr;36(2):76-81. PMID 3644262
- [Background] Neff, K. (2003). Self-Compassion: An Alternative Conceptualization of a Healthy Attitude Toward Oneself. Self and Identity, 2(2), 85-101. https://doi.org/10.1080/15298860309032